CLINICAL TRIAL: NCT03478384
Title: Pilot Study: Individualized Self-efficacy Coaching, Quality of Life and Compliance for Women With High-risk Early Breast Cancer
Brief Title: Self-efficacy Coaching for Women With Breast Cancer
Acronym: SECOM-PSWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stiftung Patientenkompetenz (Other)
Collaborators: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iOM-110393
Record Dates: First submitted 2018-03-09; First posted 2018-03-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: self-efficacy expectation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment of patients to two groups (group A: patients receive self-efficacy coaching, group B: patients do not receive additional coaching)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaching group (Experimental): Patient coaching
  Interventions: Behavioral: Patient coaching
- Control group (No Intervention): Control group - no additional coaching provided

INTERVENTIONS:
Behavioral: Patient coaching — Patients receive regular coaching to test if the coaching alters their perceived self-efficacy.
  Arms: Coaching group

SUMMARY:
This is an open, prospective, multi-center, interventional study to evaluate the benefit and efficacy of individualized self-efficacy coaching for women with high-risk early breast cancer.

In total, 6 sites will be assigned 1:1 to either the experimental arm (Group A) or the control arm (Group B). The controlled site assignment will assure a balanced site-specific QoL between both groups at baseline. All patients will be medically treated according to guidelines. The experimental Group A will in addition receive regular self-efficacy coaching.

DETAILED DESCRIPTION:
Breast cancer represents the leading cause of cancer in women in Switzerland with around 6,000 newly diagnosed cases per year. Beside the therapy- and cancer-associated somatic illness, about one third of patients develop anxiety disorders or depression and need psychotherapeutic or psychiatric care. Women with breast cancer display the highest psychic comorbidity compared to patients with other cancer entities (40% point prevalence) .

To assist with psychological coping with the disease several psycho-oncological interventions have been established in the past decades.

Self-efficacy describes the extent or strength of one's belief in one's own ability to complete tasks and reach goals. Nagel & Schreiber have developed an individualized self-efficacy coaching for cancer patients to mobilize and strengthen the belief in one's own ability to deal with and fight the disease. The SECOM-PSWE study evaluates the impact of regular self-efficacy coaching on the perceived self-efficacy and the quality of life (QoL) in patients with early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent
2. Histologically confirmed early breast cancer
3. High risk patients, defined as T≥3 and/or N+ and/or G3 and/or Triple-Negative Breast Cancer (TNBC; PgR-/ER-/HER2-) at primary diagnosis
4. Eligible for systemic neo-adjuvant or adjuvant therapy
5. Age ≥ 18 years
6. ECOG 0-2
7. Expected follow-up care at site for at least 5 years
8. Expected adherence to observation and questionnaire assessment (Group A and B) as well as to study intervention (Group A)
9. Anti-cancer therapy and follow-up care according to the established guidelines
10. Fluent in written and spoken German language

Exclusion Criteria:

1. Not eligible for systemic neo-adjuvant or adjuvant treatment according to the established guidelines
2. Previous systemic anti-neoplastic therapy
3. Resection >R0 for adjuvant patients
4. Metastases
5. Patients who decline systemic therapy according to established guidelines for personal reasons
6. Inflammatory breast cancer, sarcomas, M. Paget
7. Presence of other primary tumors within the last 5 years, except for appropriately treated, controlled, basal-cell carcinoma and cervical cancer in situ
8. Not controlled, severe, life-threatening, or prognostic unfavorable comorbidities
9. Pregnancy, lactation
10. Indication of a severe depression/anxiety disorder at baseline (PHQ 9 Score ≥15 and/or GAD-7 Score ≥15 at baseline)
11. Participation in other (non-)interventional studies or tumor registries
12. Male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Overall perceived self-efficacy | The questionnaire SWE is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Overall perceived self-efficacy is measured by a specifically developed questionnaire (questionnaire SWE). Analysis will be descriptive, separate for each group and performed according to the analysis manual. A difference between the groups is defined as 10% difference in median between the groups. The scale ranges from 10 to 40 points. The higher the score, the higher is perceived self-efficacy of the patient.

SECONDARY OUTCOMES:
Overall quality of life | The questionnaire FACT-G is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Overall quality of life is measured by the questionnaire FACT-G. Differences between the groups will be determined comparing total score. The scale ranges from 0 to 108 points. The higher the score, the better is quality of life.
Disease-related quality of life | The questionnaire FACT-B is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Disease-related quality of life is measured by the questionnaire FACT-B. Differences between the groups will be determined comparing total score. The scale ranges from 0 to 148 points. The higher the score, the better is quality of life.
Active coping with the disease | The questionnaire FKV-15 is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Active coping with the disease is measured by the questionnaire FKV-15. Differences between the groups will be determined comparing total score. The scale ranges from 15 to 75 points. The higher the score, the better the patient is coping.
Physical activity | The questionnaire IPAQ is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Physical activity is measured by the questionnaire IPAQ. Differences between the groups will be determined comparing the level of physical activity. Analysis will be done according to the scoring manual. There is no minimum or maximum for the scale, the outcome is a continuous measure presented in Metabolic Equivalent of Task (MET)-minutes. The higher the outcome, the higher is the level of physical activity.
Duration of hormone therapy | The questionnaire Compliance is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Duration of hormone therapy is determined by the questionnaire Compliance which consists of two items. Total duration of hormone therapy is measured in months and is compared between the groups. The questionnaire Compliance only applies to patients who receive hormone therapy.
Anxiety levels | The questionnaire GAD-7 is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Anxiety levels are measured by the questionnaire GAD-7. Analysis will be done according to the scoring manual. Differences between the groups will be determined comparing total score. The scale ranges from 0 to 21 points. The higher the score, the higher the level of anxiety.
Use of complementary medicine | The questionnaire I-CAM-G is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Use of complementary medicine is measured by the questionnaire I-CAM-G. The number of complementary medical measures is determined descriptively and compared between the groups.
Rate of Relapse | Occurrence of relapse is assessed at the timepoint of relapse or at 7.5 months, whichever comes first.
  Occurrence of relapse is documented during the course of the study. The occurence of relapse is assessed by the investigator as per clinical routine and documented in the eCRF by three items.
Change of perceived self-efficacy | The questionnaire SWE is collected at baseline, after 1.5 months, 4.5 months and at the timepoint of relapse or latest after 7.5 months.
  Change of perceived self-efficacy is measured by a specifically developed questionnaire (questionnaire SWE) and compared between the groups. An increase in perceived self-efficacy is defined as the first increase in total score of five or more points. The scale ranges from 10 to 40 points. The higher the score, the higher is perceived self-efficacy of the patient.
Change of quality of life | The questionnaire FACT-G is collected at baseline, after 1.5 months, 4.5 months and at the timepoint of relapse or latest after 7.5 months.
  Change of quality of life is measured by the questionnaire FACT-G and compared between the groups. An increase in quality of life is defined as the first increase in total score of five or more points. The scale ranges from 0 to 108 points. The higher the score, the better is quality of life.
Change of disease-related quality of life | The questionnaire FACT-B is collected at baseline, after 1.5 months, 4.5 months and at the timepoint of relapse or latest after 7.5 months.
  Change of disease-related quality of life is measured by the questionnaire FACT-B and compared between the groups. An increase in disease related quality of life is defined as the first increase in total score of five or more points. The scale ranges from 0 to 148 points. The higher the score, the better is quality of life.
Depression | The questionnaire PHQ-9 is collected at the timepoint of relapse or latest after 7.5 months, whichever comes first.
  Depression is measured by the questionnaire PHQ-9. Differences between the groups will be determined comparing total score. Analysis will be done according to the scoring manual. The scale ranges from 0 to 27 points. The higher the score, the higher the level of depression.
Use of micronutrients | The questionnaire I-CAM-G is collected at the timepoint of relapse or after 7.5 months, whichever comes first.
  Use of micronutrients is measured by the questionnaire I-CAM-G. The number of different types of micronutrients is determined descriptively and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Nagel, Professor MD, Study Director — Stiftung Patientenkompetenz
Locations (6):
- Switzerland (6):
  - Tumorzentrum ZeTuP Rapperswil-Jona, Rapperswil-Jona, Canton of St. Gallen
  - Prolindo, Onkologie & Hämatologie, Team am Lindenhofspital, Bern
  - Spital Thurgau AG - Kantonsspital Frauenfeld, Frauenfeld
  - Hirslanden Klinik St. Anna, Lucerne
  - Tumor-und Brustzentrum ZeTuP AG St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No